CLINICAL TRIAL: NCT03382093
Title: Personalized Feedback for Smokers With Elevated Anxiety Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lorra Garey, Clinical Psychology Doctoral Student, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR00000267; 5F31DA043390-02 (NIH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-22 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Anxiety Disorders; Anxiety; Tobacco Dependence; Smoking, Cigarette; Smoking, Tobacco
Keywords: Anxiety Sensitivity; Tobacco; Smoking; Anxiety; Feedback; Stress
MeSH Terms: conditions — Anxiety Disorders; Tobacco Use Disorder; Cigarette Smoking; Tobacco Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: If participant meets eligibility criteria, the participant will be randomly assigned to complete a computer-delivered intervention: either the (a) Personalized Feedback Intervention or (b) smoking information control.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Feedback Intervention (Active Comparator): A brief, personalized computer-delivered transdiagnostic intervention (PFI) that addresses smoking and anxiety sensitivity (AS) to reduce smoking, increase quit attempts, reduce perceived barriers to cessation, reduce AS and negative affective symptoms, and increase adaptive coping skills.
  Interventions: Behavioral: Personalized Feedback Intervention
- Smoking Information Control (Active Comparator): Standard, computer-delivered smoking cessation treatment/information.
  Interventions: Behavioral: Smoking Information Control

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — Personalized Feedback Intervention for smoking and anxiety.
  Other Names: PFI
  Arms: Personalized Feedback Intervention
Behavioral: Smoking Information Control — Smoking Information with no personalized feedback.
  Other Names: Control; Clearing the Air Pamphlet
  Arms: Smoking Information Control

SUMMARY:
This project will develop and refine a computer-delivered integrated Personalized Feedback Intervention (PFI) that directly addresses smoking and anxiety sensitivity (AS). The PFI will focus on feedback about smoking behavior, AS, and adaptive coping strategies.

DETAILED DESCRIPTION:
The primary goal of the research study is to investigate the efficacy of a brief, personalized computer-delivered transdiagnostic intervention (PFI) that addresses smoking and anxiety sensitivity (AS) to reduce smoking, increase quit attempts, reduce perceived barriers to cessation, reduce AS and negative affective symptoms, and increase adaptive coping skills compared to a smoking information only control. To address this aim, we will implement a randomized controlled trial that will employ a longitudinal experimental design and involve three stages: (a) phone-screener (pre-screener); (b) baseline appointment consisting of a pre-intervention assessment (eligibility), random assignment to a one-session computer-delivered intervention (PFI versus smoking information control with no personalized feedback), and a post-intervention assessment; (c) 1-month follow-up. Assessments will include a multi-method approach, including biological, behavioral, and self-report methods.

ELIGIBILITY:
Inclusion Criteria:

* Elevated anxiety sensitivity defined as an ASI-III score of at least 17
* Daily smoking for at least one year (minimum of 5 cigarettes per day and biochemically confirmed via Carbon Monoxide [CO] analysis at least 4 ppm)
* Not presently engaged in a quit attempt
* Not currently engaged in mental health treatment
* Capable of providing informed consent
* Willing to attend all study visits and comply with the protocol

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Students for whom you have direct access to/influence on grades
* Use of other tobacco products
* Currently suicidal or high suicide risk
* Currently psychotic or high psychotic risk
* Insufficient command of English to participate in assessment or treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate PFI | Assessed at 1-month follow-up after the one-session intervention
  Evaluate the protocol for a brief personalized, computer-delivered intervention. Assessed by program evaluation survey.

SECONDARY OUTCOMES:
Smoking Motivational Processes | Assessed at 1-month follow-up after the one-session intervention
  Smokers in intervention, relative to a smoking information control, will report increased motivation and confidence for quitting smoking. Assessed using Smoking Rulers for Change measure.
Smoking Behavior | Assessed at 1-month follow-up after the one-session intervention
  Smokers in intervention, relative to a smoking information control, will report reduced smoking rates. Assessed using Carbon Monoxide [CO] analysis.
Affective Processes | Assessed at 1-month follow-up after the one-session intervention
  Smokers in intervention, relative to a smoking information control, will report greater reductions in anxiety sensitivity. Assessed using Anxiety Sensitivity Index measure.
Mechanisms | Assessed at 1-month follow-up after the one-session intervention
  Smokers in the intervention, relative to the smoking information control, will report decreased positive consequences for continued smoking. Assessed using Smoking Consequence Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lorra L. Garey, MA, Principal Investigator — University of Houston; Michael J. Zvolensky, PHD, Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Laboratory and Substance Use Treatment Clinic, University of Houston, Houston, Texas, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03382093/Prot_SAP_000.pdf